CLINICAL TRIAL: NCT03930186
Title: A Phase 3b, Open-label, Single-arm Study of the Efficacy and Safety of Apremilast, in Subjects With Plaque Psoriasis That is Not Adequately Controlled by Topical Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-023; U1111-1230-7468 (Registry Identifier: WHO); 20200062 (Other: Amgen Study ID)
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apremilast (Experimental): After a 5-day titration, participants received 30 mg apremilast tablets orally twice daily (BID) for up to 32 weeks in addition to their existing topical therapy. At week 16 participants were permitted to decrease their use of topical therapy at their own discretion under the direction of their physician.
  Interventions: Drug: Apremilast; Drug: Topical Therapy

INTERVENTIONS:
Drug: Apremilast — Tablets for oral administration
  Other Names: CC-10004; Otezla®
Drug: Topical Therapy — Participants continued to use their existing topical treatment for psoriasis for the first 16 weeks. After 16 weeks, participants could decrease the use of topical therapy at their discretion under the direction of their physician.

SUMMARY:
The primary objective of the study is to assess the efficacy and safety of the combination of apremilast plus topical therapies for the treatment of adults with plaque psoriasis who have not achieved an adequate response with topicals alone.

DETAILED DESCRIPTION:
Participants will be enrolled at 28 sites in Japan. The study consists of 4 phases: a screening phase (4 weeks), an open-label combination therapy phase (16 weeks), an open-label combination therapy phase with optional topical reduction (16 weeks), and a post-treatment observational follow-up phase (4 weeks).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 20 years of age at the time of signing the informed consent form (ICF) with plaque psoriasis.
2. Subject has understood and voluntarily signed an informed consent document prior to any study related assessments/procedures being conducted.
3. Subject is able to adhere to the study visit schedule and other protocol requirements.
4. Subject has chronic plaque psoriasis based on a diagnosis for at least 6 months prior to Baseline.
5. Subject has psoriasis with sPGA = 2 or 3 at screening and baseline.
6. Subject is currently treated for psoriasis with topical therapies only for at least 4 weeks prior to Baseline.
7. Subject has inadequate response to current topical therapy as per Investigator's discretion.
8. Subject is naïve to all biologic therapies for psoriasis vulgaris.
9. Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination, and clinical laboratories.

   (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
10. Subjects that are females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device; tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any condition, including other inflammatory diseases or dermatologic conditions, which confounds the ability to interpret data from the study, including other types of psoriasis (ie, pustular, inverse, erythrodermic, or guttate), other than plaque psoriasis.
2. Subject has psoriatic arthritis that requires systemic therapy.
3. Subject has history of drug-induced psoriasis.
4. Subject has had prior treatment with biologic therapies for psoriasis.
5. Subject has used phototherapy or conventional systemic therapy for psoriasis within 8 weeks prior to baseline and during the study (including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine).
6. Subject has worsening of psoriasis indicated by an increase in sPGA of ≥ 1 from Screening to Baseline.
7. Subject cannot avoid excessive sun exposure or use of tanning booths for at least 8 weeks prior to Baseline and during the study.
8. Subject is currently enrolled in any other clinical trial involving an investigational product.
9. Subject has other than psoriasis, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
10. Subject has malignancy or history of malignancy or myeloproliferative or lymphoproliferative disease within the past 3 years, except for treated (ie, cured) basal cell or squamous cell in situ skin carcinomas.
11. Subject has received a live vaccine within 3 months of baseline or plans to do so during study.
12. Subject is pregnant or breastfeeding (lactating) women.
13. Subject has bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed and the infection cured, at least 4 weeks prior to Screening and no new or recurrent infections prior to the Baseline Visit.
14. Subject is hepatitis B surface antigen positive or hepatitis B core antibody positive at screening.
15. Subject is positive for antibodies to hepatitis C at screening.
16. Subject has any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
17. Subject has prior history of suicide attempt at any time in the subject's life time prior to signing the informed consent and enrollment, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.
18. Subject has active substance abuse or a history of substance abuse within 6 months prior to signing the informed consent.
19. Subject has prior treatment with apremilast or participation in a clinical study involving apremilast.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (51):
- Research Site, Erlangen, Germany
- Japan (50):
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Fukuoka-shi, Fukuoka, Fukuoka
  - Research Site, Obihiro-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sakai-shi, Osaka
  - Research Site, Bunkyo-ku, Tokyo
  - Motomachi Dermatology Clinic, Asahikawa-shi, Hokkaido
  - Research Site, Asahikawa-shi, Hokkaido
  - Nippon Medical School Hospital, Bunkyō City
  - The University of Tokyo Hospital, Bunkyō City
  - Chitose Dermatology and Plastic, Reconstructive Surgery Clinic, Chitose
  - Research Site, Chitose
  - Kiryu Dermatology Clinic, Fukuoka-shi, Fukuoka
  - Fukuoka University Hospital, Fukuoka-shi, Fukuoka
  - Tomoko Matsuda Dermatology Clinic, Fukuoka-shi, Fukuoka
  - Hino Dermatology Clinic, Fukutsu
  - Research Site, Fukutsu
  - Research Site, Kagoshima
  - Saruwatari Dermatology Clinic, Kagoshima
  - Noguchi Dermatorogy Clinic, Kamimashiki-gun
  - Research Site, Kamimashiki-gun
  - Japan Community Health-care Organization Kyushu Hospital, Kitakyushu
  - Research Site, Kitakyushu
  - Maruyama Dermatology Clinic, Koto-ku, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Mita Dermatology Clinic, Minatoku
  - Research Site, Minatoku
  - Iwate Medical University Uchimaru Medical Center, Morioka
  - Research Site, Morioka
  - Research Site, Neyagawa
  - Yoshioka Dermatology Clinic, Neyagawa
  - Takagi Dermatological Clinic, Obihiro
  - Nippon Life Hospital, Osaka
  - Research Site, Osaka
  - Hino Clinic, Sakai
  - Research Site, Sakai
  - Kume Clinic, Sakai-shi, Osaka
  - Kitagou Dermatology Clinic, Sapporo
  - Research Site, Sapporo
  - Kobayashi Skin Clinic, Sapporo
  - Hosui Medical Clinic, Sapporo
  - Sapporo Skin Clinic, Sapporo-shi, Hokkaido
  - Fukuzumi Dermatology Clinic, Sapporo-shi, Hokkaido
  - Jichi Medical University Hospital, Shimotsuke
  - Research Site, Shimotsuke
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Research Site, Shinjyuku-ku
  - Tokyo Medical University Hospital, Shinjyuku-ku
  - Fujita Health University Hospital, Toyoake
  - Research Site, Toyoake

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Abe M, Okubo Y, Takahashi H, Endo K, Chaudhari S, Deignan C, Amouzadeh H, Hino R. Consistent Efficacy of Apremilast in Patients with Psoriasis Regardless of Baseline Disease Severity or Special Area Involvement: Subgroup Analysis from PROMINENT. Dermatol Ther (Heidelb). 2024 Jun;14(6):1587-1597. doi: 10.1007/s13555-024-01179-z. Epub 2024 May 27. PMID 38801606
- [Derived] Okubo Y, Takahashi H, Hino R, Endo K, Kikuchi S, Ozeki Y, Nakamura T, Paris M, Abe M. Efficacy and Safety of Apremilast in the Treatment of Patients with Mild-to-Moderate Psoriasis in Japan: Results from PROMINENT, A Phase 3b, Open-Label, Single-Arm Study. Dermatol Ther (Heidelb). 2022 Jun;12(6):1469-1480. doi: 10.1007/s13555-022-00747-5. Epub 2022 Jun 11. PMID 35689737
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 28 centers in Japan.
Groups:
- Apremilast: Participants received 30 mg apremilast tablets orally twice daily (BID) for up to 32 weeks in addition to their existing topical therapy. At week 16, participants were permitted to decrease their use of topical therapy at their own discretion under the direction of their physician.
Period: Weeks 0 to 16
Arm/Group | Apremilast
Started | 152
Received Study Drug | 152
Completed | 140
Not Completed | 12
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 6
Period: Weeks 16 to 32
Arm/Group | Apremilast
Started | 140
Completed | 136
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (11.90)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 137
  ≥ 65 to < 75 years | 14
  ≥ 75 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 152
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: years] | 11.94 (10.629)
Body Surface Area (BSA) Affected by Psoriasis [Mean (Standard Deviation); unit: percentage of total body surface area] — The overall body surface area affected by psoriasis was estimated based on the palm area of the participant's hand, which equates to approximately 1% of total body surface area.
  BSA affected by psoriasis is expressed as a percentage of total body surface area.
  percentage of total body surface area | 13.40 (11.491)
Static Physician's Global Assessment (sPGA) Score [Count of Participants; unit: Participants] — The sPGA is an assessment by the Investigator of the overall disease severity at the time of evaluation. The National Psoriasis Foundation Psoriasis Score version of a static PGA was calculated by averaging the total body erythema, induration, and desquamation scores. Erythema (E), induration (I), and desquamation (D) were scored on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The overall scores are as follows:
  0 = Clear;
  1. = Almost Clear;
  2. = Mild;
  3. = Moderate;
  4. = Severe.
  Participants
    0 (Clear) | 0
    1 (Almost Clear) | 0
    2 (Mild) | 51
    3 (Moderate) | 101
    4 (Severe) | 0
Scalp Physicians Global Assessment (ScPGA) [Count of Participants; unit: Participants] — The ScPGA assesses scalp involvement of psoriasis. The 5-point ScPGA scale ranges from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe).
  Participants
    0 (Clear) | 17
    1 (Almost Clear) | 7
    2 (Mild) | 63
    3 (Moderate) | 63
    4 (Severe) | 2
Baseline Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: scores on a scale] — The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions.
  The PASI scores range from 0 to 72, with higher scores reflecting greater disease severity.
  scores on a scale | 8.92 (5.383)
Pruritus Visual Analog Scale (VAS) Score [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate how much itch they have had due to psoriasis in the past week by placing a vertical stroke on a 100 mm line on which the left-hand boundary (0 mm) represented no itch, and the right-hand boundary (100 mm) represented worst itch imaginable. The distance from the mark to the left-hand boundary was recorded.
  mm | 37.74 (25.257)
Baseline NAPSI Score for the Target Nail [Mean (Standard Deviation); unit: scores on a scale] — One target thumb nail or fingernail representing the worst nail psoriasis involvement was selected for assessment at Baseline.
  The nail matrix was assessed for presence of any of the nail matrix features graded on a scale of 0 (none) to 4 (present in all 4 quadrants).
  The nail bed was assessed for the presence of any nail bed features on a scale from 0 (none) to 4 ( present in all quadrants).
  The sum of the nail matrix and nail bed scores is the total score and ranges from 0 to 8 (worst).
  scores on a scale | 1.53 (2.003)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: scores on a scale] — The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 (best quality of life) to 30 (worst quality of life).
  scores on a scale | 4.63 (3.902)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an sPGA Score of Clear (0) or Almost Clear (1) at Week 16
Description: The sPGA is an assessment by the Investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The National Psoriasis Foundation Psoriasis Score version of a static PGA is calculated by averaging the total body erythema, induration, and desquamation scores. The overall scores are as follows:
  0 = Clear;
  1. = Almost Clear;
  2. = Mild;
  3. = Moderate;
  4. = Severe.
  The percentage of participants with a sPGA response was estimated using a multiple imputation method from 100 imputed data sets.
Time Frame: Week 16
Population: The enrolled population; missing values through week 16 were imputed using the multiple imputation (MI) method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percentage of participants | 43.7 [35.72 to 51.66]

2. Secondary Outcome: Percentage of Participants Who Achieved an sPGA Score of Clear (0) or Almost Clear (1) at Week 32
Description: The sPGA is an assessment by the Investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The National Psoriasis Foundation Psoriasis Score version of a static PGA is calculated by averaging the total body erythema, induration, and desquamation scores. The overall scores are as follows:
  0 = Clear;
  1. = Almost Clear;
  2. = Mild;
  3. = Moderate;
  4. = Severe.
Time Frame: Week 32
Population: The enrolled population; missing values through week 32 were imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percentage of participants | 40.8 [32.98 to 48.60]

3. Secondary Outcome: Percentage of Participants Who Achieved a Scalp Physicians Global Assessment (ScPGA) Score of Clear (0) or Almost Clear (1) at Weeks 16 and 32
Description: The ScPGA assesses scalp involvement of psoriasis based on scalp plaque elevation, scaling, and erythema. The 5-point ScPGA scale ranges from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe).
Time Frame: Weeks 16 and 32
Population: The enrolled population with Baseline ScPGA Score ≥ 2; missing values were imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 128
percentage of participants
  Week 16 | 52.3 [43.69 to 61.00]
  Week 32 | 50.8 [42.12 to 59.44]

4. Secondary Outcome: Change From Baseline in Percentage of BSA Affected by Psoriasis at Weeks 16 and 32
Description: The overall body surface area affected by psoriasis was estimated based on the palm area of the participant's hand, which equates to approximately 1% of total body surface area. BSA affected by psoriasis is expressed as a percentage of total body surface area.
  A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 16 and 32
Population: The enrolled population with available data at each time point
Measure: Mean (Standard Deviation); unit: percent BSA
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percent BSA
  Week 16: number analyzed (Participants) | 145
  Week 16 | -7.86 (8.755)
  Week 32: number analyzed (Participants) | 140
  Week 32 | -8.32 (9.478)

5. Secondary Outcome: Percent Change From Baseline in Pruritus Visual Analog Scale (VAS) at Weeks 2, 16, and 32
Description: Participants were asked to indicate how much itch they have had due to psoriasis in the past week by placing a vertical stroke on a 100 mm line on which the left-hand boundary (0 mm) represented no itch, and the right-hand boundary (100 mm) represented worst itch imaginable. The distance from the mark to the left-hand boundary was recorded. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 2, 16, and 32
Population: The enrolled population with available data at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percent change
  Week 2: number analyzed (Participants) | 143
  Week 2 | -36.96 (46.474)
  Week 16: number analyzed (Participants) | 136
  Week 16 | -28.05 (118.300)
  Week 32: number analyzed (Participants) | 132
  Week 32 | -25.29 (122.113)

6. Secondary Outcome: Mean Change From Baseline in Shiratori's Pruritus Severity Score at Weeks 2, 16, and 32
Description: Shiratori's Pruritus Severity Score is a pruritus (itchiness) severity assessment tool used in Japan. Daytime and nighttime pruritus were evaluated and scored separately. Daytime pruritus was rated on a five-grade scale: 0 (absent), 1 (endurable without scratching; minimal), 2 (subsides with slight scratching; mild), 3 (subsides with considerable scratching; moderate), or 4 (not subsiding with scratching, which prompts repeated scratching; severe).
  Nighttime pruritus was rated on a five-grade scale: 0 (absent), 1 (slight itching at bedtime but not causing intentional scratching; no difficulty sleeping because of pruritus), 2 (slight itching that subsides with scratching; no difficulty sleeping because of pruritus), 3 (difficulty sleeping because of pruritus that resolves with scratching; unconscious scratching occurs during sleep), or 4 (severe difficulty sleeping due to pruritus; frequent scratching that worsens pruritus).
  A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 2, 16, and 32
Population: The enrolled population with available data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 152
units on a scale
  Daytime: Week 2 | -0.5 (0.77)
  Daytime: Week 16: number analyzed (Participants) | 145
  Daytime: Week 16 | -0.7 (0.95)
  Daytime: Week 32: number analyzed (Participants) | 140
  Daytime: Week 32 | -0.7 (0.95)
  Nighttime: Week 2 | -0.4 (0.85)
  Nighttime: Week 16: number analyzed (Participants) | 145
  Nighttime: Week 16 | -0.7 (0.86)
  Nighttime: Week 32: number analyzed (Participants) | 140
  Nighttime: Week 32 | -0.7 (0.91)

7. Secondary Outcome: Percentage of Participants Who Achieved a ≥ 50% Reduction From Baseline in NAPSI Score (NAPSI-50) at Weeks 16 and 32 Among Participants With NAPSI ≥ 1 at Baseline
Description: One target thumb nail or fingernail representing the worst nail psoriasis involvement was selected for assessment at Baseline.
  The nail matrix was assessed for presence of any of the nail matrix features (pitting, leukonychia red spots in the lunula, crumbling) graded on a scale of 0 (none) to 4 (present in all 4 quadrants).
  The nail bed was assessed for the presence of any nail bed features (onycholysis, splinter hemorrhages, subungual hyperkeratosis, "oil drop" (salmon patch dyschroma) on a scale from 0 (none) to 4 (present in all quadrants).
  The sum of the nail matrix and nail bed scores is the total score and ranges from 0 to 8 (worst).
Time Frame: Weeks 16 and 32
Population: The enrolled population with Baseline NAPSI Score ≥ 1; missing data were imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 76
percentage of participants
  Week 16 | 44.7 [33.56 to 55.92]
  Week 32 | 57.9 [46.79 to 68.99]

8. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Weeks 16 and 32
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much), except for Question 7, which first asks whether the participant's skin prevented them from working or studying (Yes (score = 3) or No (score = 0), then If "No", the participant is asked how much their skin was a problem at work or studying over the last week, with responses from 0 (not at all), 1 (a little), or 2 (a lot).
  The DLQI total score ranges from 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 16 and 32
Population: The enrolled population with available data at each time point
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 152
scores on a scale
  Week 16: number analyzed (Participants) | 145
  Week 16 | -2.2 (2.96)
  Week 32: number analyzed (Participants) | 140
  Week 32 | -2.3 (2.97)

9. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Weeks 16 and 32
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. The PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 16 and 32
Population: The enrolled population with available data at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percent change
  Week 16: number analyzed (Participants) | 145
  Week 16 | -69.61 (22.896)
  Week 32: number analyzed (Participants) | 140
  Week 32 | -69.48 (25.421)

10. Secondary Outcome: Percentage of Participants Who Achieved ≥ 75% Reduction From Baseline in PASI Score (PASI-75)
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. The PASI scores range from 0 to 72, with higher scores reflecting greater disease severity.
Time Frame: Weeks 16 and 32
Population: The enrolled population; missing values were imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percentage of participants
  Week 16 | 43.4 [35.54 to 51.30]
  Week 32 | 46.7 [38.78 to 54.64]

11. Secondary Outcome: Percentage of Participants Who Achieved ≥ 50% Reduction From Baseline in PASI Score (PASI-50)
Description: as for outcome 10
Time Frame: Weeks 16 and 32
Population: The enrolled population; missing data was imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percentage of participants
  Week 16 | 79.6 [73.20 to 86.01]
  Week 32 | 75.0 [68.12 to 81.88]

12. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Sub-domain Scores
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) version II is a self-administered instrument to understand a participant's satisfaction on current therapy. The TSQM comprises 11 items across 4 domains focusing on effectiveness (Item 1 and 2), side effects (Item 4 to 6), convenience (Item 7 to 9), and global satisfaction (Item 10 and 11). With the exception of Item 3 (experience any side effects; yes or no), all items have five or seven responses. Item scores are summed to give four domain scores, which are in turn transformed to a scale from 0 (extremely dissatisfied) to 100 (extremely satisfied).
Time Frame: Baseline and weeks 16 and 32
Population: The enrolled population with available data at each time point
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 152
scores on a scale
  Effectiveness: Baseline | 52.25 (17.553)
  Effectiveness: Week 16: number analyzed (Participants) | 145
  Effectiveness: Week 16 | 67.41 (21.176)
  Effectiveness: Week 32: number analyzed (Participants) | 140
  Effectiveness: Week 32 | 68.93 (19.067)
  Side Effects: Baseline | 97.37 (10.078)
  Side Effects: Week 16: number analyzed (Participants) | 145
  Side Effects: Week 16 | 90.40 (17.714)
  Side Effects: Week 32: number analyzed (Participants) | 140
  Side Effects: Week 32 | 93.21 (14.947)
  Convenience: Baseline | 56.43 (16.735)
  Convenience: Week 16: number analyzed (Participants) | 145
  Convenience: Week 16 | 70.34 (17.201)
  Convenience: Week 32: number analyzed (Participants) | 140
  Convenience: Week 32 | 70.48 (16.527)
  Global Satisfaction: Baseline | 55.43 (18.554)
  Global Satisfaction: Week 16: number analyzed (Participants) | 145
  Global Satisfaction: Week 16 | 71.21 (18.241)
  Global Satisfaction: Week 32: number analyzed (Participants) | 140
  Global Satisfaction: Week 32 | 70.71 (18.660)

13. Secondary Outcome: Percentage of Participants Who Achieved a Patient Benefit Index (PBI) Score ≥ 1 at Weeks 16 and 32
Description: The Patient Benefit Index (PBI) is used to assess patient-relevant benefits of psoriasis treatment as a function of the most important needs identified by the participant before the start of treatment.
  Participants were asked to assess the benefits of treatment by completing the Patient Benefit Questionnaire (PBQ), which consists of 25 treatment goal statements scored from 0 (not at all) to 4 (very).
  The PBI is calculated for each participant by weighing the achievement values of each statement by their importance to the individual patient as assessed prior to the start of treatment. The PBI ranges from 0 (no benefit) to 4 (maximum benefit).
Time Frame: Weeks 16 and 32
Population: The enrolled population; missing data was imputed using non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
percentage of participants
  Week 16 | 91.4 [87.00 to 95.89]
  Week 32 | 88.2 [83.02 to 93.29]

14. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: The Investigator assessed the severity/intensity of each adverse event as:
  Mild (asymptomatic or mild symptoms; intervention not indicated; activities of daily life (ADLs) minimally or not affected); Moderate (symptom(s) cause moderate discomfort; local or noninvasive intervention indicated; more than minimal interference with ADLs but able to carry out daily social and functional activities; drug therapy may be required); Severe (symptoms causing severe discomfort/pain; symptoms requiring medical/surgical attention/intervention; interference with ADLs including inability to perform daily social and functional activities; drug therapy required).
  A serious adverse event is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event.
Time Frame: From first dose of study drug until at least 28 days after last dose; up to 36 weeks.
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 152
Participants
  Any treatment-emergent adverse event | 115
  Drug-related TEAE | 88
  Severe TEAE | 4
  Serious TEAE | 4
  Severe drug-related TEAE | 1
  Serious drug-related TEAE | 1
  TEAE leading to drug interruption | 3
  TEAE leading to drug withdrawal | 7
  TEAE leading to death | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until at least 28 days after last dose; up to 36 weeks.
Groups:
- Apremilast 30 mg: Participants received 30 mg apremilast tablets orally twice daily (BID) for up to 32 weeks in addition to their existing topical therapy. At week 16, participants were permitted to decrease their use of topical therapy at their own discretion under the direction of their physician.
Arm/Group | Apremilast 30 mg
All-Cause Mortality (participants affected / at risk) | 0/152
Serious Adverse Events (participants affected / at risk) | 4/152
Other Adverse Events (participants affected / at risk) | 84/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast 30 mg (N=152)
Deafness unilateral (Ear and labyrinth disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast 30 mg (N=152)
Diarrhoea (Gastrointestinal disorders) | 29
Faeces soft (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 29
Nasopharyngitis (Infections and infestations) | 28
Headache (Nervous system disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03930186/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03930186/SAP_001.pdf